CLINICAL TRIAL: NCT01331850
Title: A Randomized Open-label Study to Evaluate the Sustained Virologic Response of Danoprevir/Ritonavir and Copegus in Combination With RO5024048 and/or Pegasys in Chronic Hepatitis C Genotype 1 Patients Who Failed Previous Standard Therapy
Brief Title: A Study of Danoprevir/Ritonavir and Copegus With RO5024048 and/or Pegasys in Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WV21913; 2010-019585-90
Record Dates: First submitted 2011-03-28; First posted 2011-04-08 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a; danoprevir; Ritonavir

ARMS (6):
- Previous null responders (Cohort B): Group 4 (Experimental): Patients in all groups will receive danoprevir 100 mg twice a day and ritonavir 100 mg twice a day for 24 weeks. In addition, Group 4 will receive RO5024048 1000 mg twice a day and Copegus 1000 mg or 1200 mg twice a day for 24 weeks.
  Interventions: Drug: Copegus; Drug: RO5024048; Drug: danoprevir; Drug: ritonavir
- Previous null responders (Cohort B): Group 5 (Experimental): Patients in all groups will receive danoprevir 100 mg twice a day and ritonavir 100 mg twice a day for 24 weeks. Group 5 will receive RO5024048 1000 mg twice a day, Pegasys 180 microgram subcutaneously once weekly and Copegus 1000 mg or 1200 mg twice a day for 24 weeks.
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: RO5024048; Drug: danoprevir; Drug: ritonavir
- Previous null responders (Cohort B): Group 6 (Experimental): Patients in all groups will receive danoprevir 100 mg twice a day and ritonavir 100 mg twice a day for 24 weeks. Group 6 will receive RO5024048 1000 mg twice a day, Pegasys 180 microgram subcutaneously once weekly and Copegus 1000 mg or 1200 mg twice a day for 24 weeks. In addition, patients in Group 6 will receive another 24 weeks of Pegasys plus Copegus treatment.
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: RO5024048; Drug: danoprevir; Drug: ritonavir
- Previous partial responders (Cohort A): Group 1 (Experimental): Patients in all groups will receive danoprevir 100 mg twice a day and ritonavir 100 mg twice a day for 24 weeks. In addition, Group 1 will receive RO5024048 1000 mg twice a day and Copegus 1000 mg or 1200 mg twice a day for 24 weeks.
  Interventions: Drug: Copegus; Drug: RO5024048; Drug: danoprevir; Drug: ritonavir
- Previous partial responders (Cohort A): Group 2 (Experimental): Patients in all groups will receive danoprevir 100 mg twice a day and ritonavir 100 mg twice a day for 24 weeks. In addition, Group 2 will receive Pegasys 180 microgram subcutaneously once weekly and Copegus 1000 mg or 1200 mg twice a day for 24 weeks.
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: danoprevir; Drug: ritonavir
- Previous partial responders (Cohort A): Group 3 (Experimental): Patients in all groups will receive danoprevir 100 mg twice a day and ritonavir 100 mg twice a day for 24 weeks. Group 3 will receive RO5024048 1000 mg twice a day, Pegasys 180 microgram subcutaneously once weekly and Copegus 1000 mg or 1200 mg twice a day for 24 weeks.
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: RO5024048; Drug: danoprevir; Drug: ritonavir

INTERVENTIONS:
Drug: Copegus — 1000 mg or 1200 mg daily oral doses for 24 weeks
  Arms: Previous null responders (Cohort B): Group 4; Previous null responders (Cohort B): Group 5; Previous partial responders (Cohort A): Group 1; Previous partial responders (Cohort A): Group 2; Previous partial responders (Cohort A): Group 3
Drug: Copegus — 1000 mg or 1200 mg daily oral doses for 48 weeks
  Arms: Previous null responders (Cohort B): Group 6
Drug: Pegasys — 180 microgram subcutaneously once weekly for 24 weeks
  Arms: Previous null responders (Cohort B): Group 5; Previous partial responders (Cohort A): Group 2; Previous partial responders (Cohort A): Group 3
Drug: Pegasys — 180 microgram subcutaneously once weekly for 48 weeks
  Arms: Previous null responders (Cohort B): Group 6
Drug: RO5024048 — 1000 mg oral doses twice a day for 24 weeks
  Arms: Previous null responders (Cohort B): Group 4; Previous null responders (Cohort B): Group 5; Previous null responders (Cohort B): Group 6; Previous partial responders (Cohort A): Group 1; Previous partial responders (Cohort A): Group 3
Drug: danoprevir — 100 mg oral doses twice a day for 24 weeks
Drug: ritonavir — 100 mg oral doses twice a day for 24 weeks

SUMMARY:
This randomized, open-label, multi-center study will evaluate the sustained virological response, pharmacokinetics and safety of various combinations of danoprevir/ritonavir with Copegus plus RO5024048 and/or Pegasys in patients with chronic hepatitis C infection. Patients will be divided into 2 separate cohorts. Cohort A, previous partial responders, will be randomized to Groups 1-3 and cohort B, previous null responders, will be randomized to Groups 4-6. Patients in all groups will receive danoprevir 100 mg twice a day and ritonavir 100 mg twice a day for 24 weeks. In addition, Groups 1 and 4 will receive RO5024048 1000 mg twice a day and Copegus 1000 mg or 1200 mg twice a day for 24 weeks; Group 2 will receive Pegasys 180 microgram subcutaneously once weekly and Copegus 1000 mg or 1200 mg twice a day for 24 weeks; Groups 3, 5 and 6 will receive RO5024048 1000 mg twice a day, Pegasys 180 microgram subcutaneously once weekly and Copegus 1000 mg or 1200 mg twice a day for 24 weeks. In addition, patients in Group 6 will receive another 24 weeks of Pegasys plus Copegus treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, age 18 years and older
* Presence of hepatitis C infection, genotype 1a or 1b
* Documentation of previous treatment failure after receiving approved doses of peginterferon plus ribavirin for at least 12 weeks
* Patients must have discontinued prior hepatitis C treatment at least 12 weeks prior to study start

Exclusion Criteria:

* Infection with any hepatitis C genotype or subtype other than genotype 1a or 1b
* Patients with cirrhosis
* Patients who were discontinued from previous peginterferon plus ribavirin therapy due to reasons other than insufficient therapeutic response
* Co-infection with hepatitis B or human immunodeficiency virus (HIV)
* History or evidence of chronic liver disease other than hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Sustained virological response (SVR) of danoprevir/ritonavir with RO5024048 and Copegus in patients with previous partial or null response to peginterferon/ribavirin treatment | 24 weeks
Sustained virological response (SVR) of danoprevir/ritonavir with Pegasys and Copegus in patients with previous partial response to peginterferon/ribavirin treatment | 24 weeks
Sustained virological response (SVR) of danoprevir/ritonavir and RO5024048 with Pegasys and Copegus in patients with previous partial or null response to peginterferon/ribavirin treatment | 24 weeks
Sustained virological response (SVR) of danoprevir/ritonavir and RO5024048 with Pegasys and Copegus followed by 24 weeks of Pegasys and Copegus treatment in patients with previous null response to peginterferon/ribavirin treatment | 48 weeks

SECONDARY OUTCOMES:
Safety (Incidence of adverse events) of danoprevir, RO5024048 and Copegus | 48 weeks
Safety (Incidence of adverse events) of danoprevir, Pegasys and Copegus | 48 weeks
Safety (Incidence of adverse events) of danoprevir, RO5024048, Pegasys and Copegus | 72 weeks
Virological response over time | 48 weeks
Change in danoprevir plasma concentration | 24 weeks
Change in RO5024048 plasma concentration | 24 weeks
Hepatitis C virus drug resistance profile | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (59):
- United States (18):
  - La Jolla, California
  - Long Beach, California
  - Sacramento, California
  - San Diego, California
  - Aurora, Colorado
  - Orlando, Florida
  - Decatur, Georgia
  - Chicago, Illinois
  - New Orleans, Louisiana
  - Detroit, Michigan
  - Manhasset, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Medford, Oregon
  - Providence, Rhode Island
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
- Australia (5):
  - Darlinghurst, New South Wales
  - Kingswood, New South Wales
  - Westmead, New South Wales
  - Adelaide, South Australia
  - Melbourne, Victoria
- Vienna, Austria
- Brazil (2):
  - Porto Alegre, Rio Grande do Sul
  - Ribeirão Preto, São Paulo
- Canada (6):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
- France (4):
  - La Tronche
  - Paris
  - Pessac
  - Vandœuvre-lès-Nancy
- Germany (4):
  - Berlin
  - Essen
  - Kiel
  - Tübingen
- Italy (4):
  - Napoli, Campania
  - Milan, Lombardy
  - Pavia, Lombardy
  - Pisa, Tuscany
- Guadalajara, Mexico
- Poland (5):
  - Bydgoszcz
  - Czeladź
  - Kielce
  - Lodz
  - Warsaw
- San Juan, Puerto Rico
- Spain (4):
  - Badalona, Barcelona
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Seville, Sevilla
- United Kingdom (4):
  - Birmingham
  - Dundee
  - London
  - Manchester